CLINICAL TRIAL: NCT02851043
Title: Non-Invasive Respiratory Monitor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Tariq Rahman, Principal Research Engineer, Nemours Children's Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 613308
Record Dates: First submitted 2016-07-19; First posted 2016-08-01 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neuromuscular Diseases; Healthy Volunteers
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pneuRIP(breathing with resistance) (Experimental): Testing the subjects breathing with resistance
  Interventions: Device: pneuRIP (breathing with resistance); Device: Respitrace system (Carefusion) (breathing without resistance)
- Respitrace system (Carefusion) (breathing without resistance) (No Intervention): Testing subjects breathing without resistance

INTERVENTIONS:
Device: pneuRIP (breathing with resistance) — subjects are given a resistance element to breath through
  Arms: pneuRIP(breathing with resistance)
Device: Respitrace system (Carefusion) (breathing without resistance) — subjects are asked to breath normally
  Arms: pneuRIP(breathing with resistance)

SUMMARY:
This study will clinically evaluate a newly developed respiratory monitor - pneuRIP. The pneuRIP uses Respiratory Inductance Plethysmography (RIP) bands to measure key breathing indices non-invasively. This study compares the pneuRIP to an existing Respitrace system (Carefusion, Yorba Linda CA). 10 normal children and 10 children with breathing difficulties will be monitored with both systems.

DETAILED DESCRIPTION:
Firstly, ten healthy children will participate in a trial to evaluate the pneuRIP. They will be fitted with the bands around their abdomen and chest. The pneuRIP will be connected to the bands through electrodes. Breathing is then measured wirelessly with an iPad. They will be asked to lie down. They are asked to breath normally then asked to breath with a resistive elements to place in their mouth. The resistive elements makes it difficult to breath (similar to breathing through a straw). They will breathe for 3 minutes for both conditions as we record their breathing with the pneuRIP and the Respitrace. These data will be compared.

Secondly, A group of 10 subjects from the outpatient muscle clinic will be fitted with the chest and abdomen bands. The Respitrace monitor and the pneuRIP will record their breathing patterns. Data from the two systems will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Neuromuscular disease subjects with mild breathing difficulty
* Capable of following verbal instructions

Exclusion Criteria:

* Severe breathing difficulties

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Breathing rate | Immediately after test
  The breathing rate is measured by two different monitors

SECONDARY OUTCOMES:
Labored breathing Index | Immediately after test
  The labored breathing index is measured by two different monitors
Phase Difference | Immediately after test
  The phase difference between the pneuRIP and Respitrace is measured by two different monitors
Percent rib cage | Immediately after test
  The percentage of breathing performed by the rib cage is measured by two different monitors

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Shaffer, PhD, Principal Investigator — Nemours
Locations (1):
- Nemours/A.I. duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No